CLINICAL TRIAL: NCT02148926
Title: Clinical and Genetic Examinations of Dilated Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Morris Hey, MD, Phd. student, University of Southern Denmark
Other Study IDs: DCM-011213-28037
Record Dates: First submitted 2014-05-23; First posted 2014-05-29 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA for genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a descriptive study to investigate clinical and genetic features of dilated cardiomyopathy (DCM) patients and their relatives. 109 probands with DCM have been clinically characterized with clinical examinations including ECG and echocardiography, and furthermore they have had next generation sequencing (NGS) of 42 known DCM genes, and 34 candidate genes. The probands were consequtively included in the study and 59 had undergone heart transplantation (HTx) upon inclusion. of these patients underwent heart transplantation. The data from NGS is validated by Sanger sequencing. In this study we will examine the relatives to the 109 index patients by genetic and clinical cascade screening including advanced echocardiography including 3D volume measurements and speckle-tracking (GLS). Genetic investigations of relatives will be performed if a disease-associated mutation is identifed in the proband. Approximately 480 clinical examinations will be performed this way to be able to:

1a. Investigate the frequency of familial types of DCM

1b. To investigate the yield of genetic and clinical cascade screening

2. To describe genotype phenotype correlations

3. To investigate if there are subtle changes in the heart in genopositive individuals which do not meet the conventional diagnostic criteria evaluated by advanced echocardiography.

DETAILED DESCRIPTION:
Title:

Clinical and genetic examinations of dilated cardiomyopathy

Background:

Dilated cardiomyopathy (DCM) is a severe disease of the heart muscle characterised by reduced pumping function and dilatation of the left ventricle without any obvious cause like hypertension, ischemic heart disease or heart valve disease. The patients often complain about shortness of breath, oedemas, and fatigability. The first sign of the disease can be a severe heart rhythm disorder without any preceding symptoms and DCM is not a rare cause of suddenly unexpected death. DCM is a frequent reason for heart transplantation and the prognosis is severe though improved over the last decades with the implementation of modern heart failure treatment.

The prevalence of DCM is around 1:2500 in the vestern world and multiple screening studies of first generation relatives to DCM patients have shown that in 30-50% of the cases it was possible to identify at least one other relative with the same disease. The inheritance is often dominant and at this point there has been reported disease associated mutations in over 40 different genes. The clinical examinations of affected families have shown that the expression of the disease varies from very critical symptoms and changes in the heart to discrete changes of the heart with no accompanying symptoms. Furthermore the time of debut of DCM can vary a lot even within the same family and the disease can manifest itself from early childhood to late adulthood.

Newer investigations indicate that a subgroup of approximately 10-15% of inherited DCM cases has a higher incidence of severe heart rhythm disorders and thereby worsened prognosis. In a considerable part of these families the disease is caused by a genetic mutation in a specific gene that codes for a nuclear membrane protein and that mutation is labelled lamin A/C. The recognition of the linkage between the genotype and the clinical presentation of the disease (phenotype), has formed the foundation of clinical algorithms and made it possible to improve the individualised risk stratification and the choice of treatment.

Status:

There is a general consensus to offer clinical screening for heart disease to relatives of younger DCM patients to be able to detect the disease before symptoms arise and if necessary commence early treatment and thus avoid serious disease complications and improve the prognosis. In families where the clinical examinations did not reveal any other relatives with signs of the disease, it is unclear if there is any benefit in continued controls of the apparently healthy relatives to reveal a possible later debut of the disease. The hope is that genetic investigations can assist in clarifying this question. If it is possible to identify a disease related genetic mutation in the index patient with DCM, it would be possible to offer genetic diagnostics to relatives and hereby identify mutation carriers in risk of developing the disease and offer these relatives relevant clinical controls and disease monitoring, while relatives without the mutation can be discharged without any further investigations.

Until recently it has not been technically and financially possible to offer routine genetic diagnostics due to large number of disease related genes and an unknown number of unidentified DCM associated genes at this point. Fortunately there has been a revolutionary development in DNA sequencing technology through the last couple of years making it possible to examine an almost unlimited amount of genes in large patient cohorts fast and to an acceptable expense. The Technology is called "Next Generation Sequencing" (NGS), and it can also be used to discover new disease associated genes and do genetic association studies.

Motivation:

The main supervisor of the project, professor Jens Mogensen has been participating in an EU financed FP7 research project called INHERITANCE (INtegrated HEart Research In TrANslational genetics and Cardiomyopathies in Europe) since 2010. The purpose of this project is to perform clinical and genetic examinations of DCM patients. The project participants comes from 11 internationally recognised European centres lead by Professor Arbustini from Pavia in Italy (www.inheriatanceproject.eu). Due to the NGS technology is has been possible to make genetic examinations on 800 European DCM patients in 42 known disease associated genes as a part of the project. Furthermore 34 candidate genes were included which from a theoretical point of view could be new disease associated genes. The Danish cohort has contributed with 140 well characterised DCM patients from Funen and Jutland.

The raw NGS data performed by the group of Professor Katus in Heidelberg, Germany is being assessed by the bioinformatics at the department of clinical genetics in Vejle and they are processing the sequencing data on the Danish patients. The first results have been processes and the final results are expected to be available in the summer of 2014.

The Danish DCM cohort is characterised by containing approximately 50% HTx patients and 50% with stable disease. This makes it possible to compare the genetic aetiology between the consecutively transplanted patients and the non transplanted patients and hereby get an impression of the relationship between prognosis and the occurrence of different mutations in certain genes.

Purpose:

1.To perform clinical and genetic investigations of DCM patients and their relatives to be able to:

1a. Investigate the frequency of familial types of DCM

1b. Investigate the yield of genetic and clinical cascade screening

2. Describe genotype phenotype correlations including possible differences in genotype among transplanted patients compared to non-transplanted.

3. Investigate if there are subtle changes in the heart in genopositive individuals which do not meet the conventional diagnostic criteria evaluated by advanced echocardiography.

Research schedule:

Clinical examinations of index patients:

Already 109 DCM probands has been included in the cohort and all data is gathered in a database.

Clinical examinations of relatives to the index patients:

1. Relatives will get a conventional clinical examination according to guidelines, an ECG and echocardiography. If it is indicated a MRI scan or invasive investigations will be performed according to clinical guidelines.
2. Conventional echocardiography: Conventional two dimensional (2D), tissue Doppler and Doppler echocardiography will be used to evaluate systolic and diastolic function of the left ventricle and the outflow tract conditions of the left ventricle (LVOT). The examinations will be performed on a Philips Epiq7 medical ultrasound machine and stored digitally for later blinded analysis. The examination will be performed according to national guidelines hence recording a parasternal long axis view with zoom of the LVOT, then a parasternal short axis view on aortic valve, mitral valve and papillary muscle level. From the apex recording a 4 chamber view, apical 2 chamber view and apical long axis view. When recording 2D, two consecutive loops are saved. Continuous wave (CW) Doppler through the aortic valve and the tricuspid valve, pulsed wave (PW) Doppler through the LVOT and of the mitral inflow is also performed. PW tissue Doppler of the lateral and medial mitral annulus is performed. When performing Doppler examinations sweep velocities at 100 mm/s is used with simultaneous ECG registration. Five consecutive heart beats are recorded and saved. Furthermore colour Doppler of the aortic-, the mitral- and the tricuspid valve is recorded to estimate the degree of regurgitation for every valve. More than a mild mitral regurgitation will be further quantified by effective regurgitation orifice (ERO).

Advanced echocardiography: Zoom of the left ventricle with frame rates of 60-100 fps recorded in apical 4 chamber, 2 chamber and apical long axis will be performed and saved for later blinded analysis with speckle tracking analysis, evaluation of torsion and twist, and global longitudinal strain (GLS). Furthermore a zoomed view of the left atrium in 4 chamber and 2 chamber views will be saved and 3 dimensional (3D) views of the left ventricle, right ventricle and left atrium will be performed.

Time schedule and milestones for the remaining clinical examinations:

It is expected that relatives to the DCM patients included will be offered the possibility to participate in this study. Experience shows that in average about 4 relatives pr index patient will be offered clinical examination, thus roughly 480 clinical examinations is still to be performed. The clinical examinations will be performed on the cardiology departments at Odense University Hospital (OUH) and Aarhus University Hospital (AUH) in collaboration with DMSc Hans Eiskjaer. The examinations are expected to be completed in September 2015. The relatives will be informed about the genetic results continuously, and they will be offered genetic counselling according to usual guidelines.

Practical preconditions for the clinical examinations to be performed:

The necessary medical expertise and the necessary medical equipment have to be available at the cardiology departments mentioned above.

Genetic examinations:

In those cases where a presumable diseas-associated mutation is identified and several family members in the same family has DCM, Sanger sequencing of the relevant family members will be undertaken. The results will be used in a coherent evaluation to estimate if there is enough evidence to classify the sequence variation as definitely disease related or as a variant of unknown importance.

Time schedule and milestones for the genetic examinations:

The final NGS sequencing results is expected to be available in the spring of 2014. Sequencing of the family members is expected to be performed simultaneously with the clinical examinations.

Practical preconditions for the genetic examinations to be performed:

The necessary molecular biological expertise and the necessary equipment have to be available at the clinical genetic department of Vejle Hospital.

Supervisors:

Primary Supervisor: Professor, DMSc, Jens Mogensen, the cardiology department of OUH Co supervisor: DMSc Jacob Moeller, the cardiology department of OUH Co supervisor: DMSc Hans Eiskjaer, the cardiology department of AUH

Ethical considerations:

It is likely that the participants in the study will benefit from the results with regards to enhanced individual counselling and risk stratification. If the participants do not wish to know of their own or their relatives genetic constitution it will be respected and considerations regarding diagnostics and treatment will follow the applicable international guidelines. It is the supervisors and the other ones responsible for the project perception that the possible benefits, outweighs the risks and side effects of this study. The project has been approved by the Committee of Health Research Ethics in central Denmark region and is furthermore approved by the Danish Data Protection Agency.

ELIGIBILITY:
Inclusion Criteria:

* Related to one of the index patients
* Available for genetic testing and clinical examinations

Exclusion Criteria:

* Death
* Not available for genetic testing and clinical examinations

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families in Denmark with history of dilated cardiomyopathy. Patients mainly from Funen and Jutland.
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Genetics | 3 years
  Difference in the genetics in the transplanted vs the non-transplanted group

SECONDARY OUTCOMES:
Global longitudinal strain | 3 years
  GLS in genopositive patients with no expression of the disease according to guidelines precipitating reduction in ejection fraction. Assesing differences in GLS in the genopositive vs the genonegative group at baseline in the individuals with no signs of DCM.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Mogensen, Professor, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided